CLINICAL TRIAL: NCT05599191
Title: A Phase 3, 52-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm Efficacy and Safety Study With Open-Label Extension of BLU-5937 in Adult Participants With Refractory Chronic Cough, Including Unexplained Chronic Cough (CALM-1)
Brief Title: A 52-Week Study of the Efficacy and Safety of BLU-5937 in Adults With Refractory Chronic Cough
Acronym: CALM-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221850; BUS-P3-01 (Other: Bellus Health Inc); 2024-513460-26-00 (Other: EU CT Number)
Record Dates: First submitted 2022-10-18; First posted 2022-10-31 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cough; Refractory Chronic Cough
Keywords: Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; Cough; Chronic Cough
MeSH Terms: conditions — Cough; Chronic Cough; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory | interventions — BLU-5937

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BLU-5937 25 mg (Experimental): BLU-5937 oral dose 25 mg twice a day.
  Interventions: Drug: BLU-5937
- BLU-5937 50 mg (Experimental): BLU-5937 oral dose 50 mg twice a day.
  Interventions: Drug: BLU-5937
- Placebo (Placebo Comparator): Matching Placebo for BLU-5937 oral dose twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLU-5937 — Oral administration of BLU-5937 Tablets
  Other Names: Camlipixant
  Arms: BLU-5937 25 mg; BLU-5937 50 mg
Drug: Placebo — Oral administration of matching placebo for BLU-5937 Tablets
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-arm, Phase 3 study of BLU-5937 in participants with Refractory Chronic Cough (RCC).

DETAILED DESCRIPTION:
The primary efficacy objective is to assess the effect of BLU-5937 on 24-hour cough frequency in adults with refractory chronic cough (including unexplained chronic cough) at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Refractory chronic cough (including unexplained chronic cough) for at least one year
* Women of child-bearing potential must use a highly effective contraception method during the study and for at least 14 days after the last dose

Exclusion Criteria:

* Current smoker/vaper (all forms of smoking and inhaled substances, including, cannabis/tobacco smoke and nicotine vapors) or individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history
* Diagnosis of chronic obstructive pulmonary disease, bronchiectasis, chronic bronchitis, cystic fibrosis, pulmonary sarcoidosis, idiopathic pulmonary fibrosis, uncontrolled asthma, or other significant or progressive airway/respiratory disorder that might affect cough based on clinician assessment
* Respiratory tract infection within 4 weeks before screening
* Laboratory confirmed Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection at screening
* History of malignancy in the last 5 years
* History of alcohol or drug abuse within the last 3 years
* Has a positive serologic test for human immunodeficiency virus (HIV), hepatitis B virus surface antigen, or hepatitis C virus.
* Previous participation in a BLU-5937 trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
24-Hour Cough Frequency | Week 12
  Assessed using an ambulatory cough monitor
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) up to Week 52 | Up to Week 52
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product and which does not necessarily have a causal relationship with that product. An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death, is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; or other situations as per the medical or scientific judgment of the Investigator.
Number of Participants with Adverse Events of Medical Interest (AEMIs) up to Week 52 | Up to Week 52
  An AEMI is an event of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring is appropriate. The following are AEMIs for this study: taste disturbance, oral hypoesthesia, oral paresthesia, and new or worsening findings of the cornea.
Number of Participants with Study Treatment Discontinuation due to AEs and SAEs up to Week 52 | Up to Week 52
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product and which does not necessarily have a causal relationship with that product. An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death, is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; or other situations as per the medical or scientific judgment of the Investigator.
Number of Participants with AEs and SAEs Leading to Study Withdrawal up to Week 52 | Up to Week 52
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product and which does not necessarily have a causal relationship with that product. An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death, is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; or other situations as per the medical or scientific judgment of the Investigator.
Change from Baseline in Vital Signs: Systolic and Diastolic Blood Pressure (millimeters of mercury [mm Hg]) at Week 52 | Baseline, Week 52
Change from Baseline in Vital Sign: Pulse (beats per minute) at Week 52 | Baseline, Week 52
Change from Baseline in Vital Sign: Respiratory Rate (breaths per minute) at Week 52 | Baseline, Week 52
Change from Baseline in Vital Sign: Body Temperature (degrees Celsius) at Week 52 | Baseline, Week 52
Change from Baseline in Vital Sign: Weight (kilograms [kg]) at Week 52 | Baseline, Week 52
Change from Baseline in Male Reproductive Hormone: Total Testosterone (nanomoles per liter [nmol/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Male Reproductive Hormones: Follicle-Stimulating Hormone [FSH] and Luteinizing Hormone [LH] (international units per liter [IU/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Male Reproductive Hormone: Inhibin B (nanograms per liter [ng/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameter: Red Blood Cell (RBC) Count (10^12 cells per liter) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameters: Hemoglobin and Mean Corpuscular Hemoglobin Concentration (MCHC) (grams per liter [g/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameter: Hematocrit (percentage) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameter: Mean Corpuscular Volume (MCV) (femtoliters [fL]) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin (MCH) (picograms per cell [pg/cell]) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameter: Red Cell Distribution Width (RDW) (percentage) at Week 52 | Baseline, Week 52
Change from Baseline in Hematology Parameters: White Blood Cell (WBC) Count (neutrophils, lymphocytes, monocytes, eosinophils, and basophils) and Platelet Count (10^9 cells per liter) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Gamma-Glutamyl Transferase (GGT) (units per liter [U/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameters: Alkaline Phosphatase (ALP) and Creatine Kinase (CK) (international units per liter [IU/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameters: Total Bilirubin, Direct and Indirect Bilirubin, and Creatinine (micromoles per liter) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameters: Sodium, Potassium, Chloride, Calcium, Magnesium, Bicarbonate, Glucose, and Blood Urea Nitrogen (BUN) (millimoles per liter [mmol/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameters: Protein and Albumin (grams per liter [g/L]) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameter: Estimated Glomerular Filtration Rate (eGFR) (milliliters per minute per 1.73 meters squared [mL/min/1.73 m^2]) at Week 52 | Baseline, Week 52
Change from Baseline in Clinical Chemistry Parameters: Prothrombin Time (PT) and Activated Partial Thromboplastin Time (aPTT) (seconds) at Week 52 | Baseline, Week 52
Change from Baseline in Electrocardiogram (ECG) Value: Heart Rate (beats per minute) at Week 52 | Baseline, Week 52
Change from Baseline in ECG Value: PR Interval, QT Interval, RR Interval, QRS Interval, and Corrected QT Interval Using Fridericia's Formula (QTcF) (milliseconds) at Week 52 | Baseline, Week 52

SECONDARY OUTCOMES:
Change from Baseline in Cough Severity Visual Analogue Scale at Week 12 | Baseline, Week 12
  Assessed by Cough Severity Visual Analogue Scale [VAS] by the participant on a 100 mm visual analogue scale where higher scores indicate greater severity.
Percentage of Participants With Greater than or Equal to (>=) 30 mm Reduction From Baseline in Cough Severity Visual Analogue Scale at Week 12 | Baseline, Week 12
  Assessed by Cough Severity Visual Analogue Scale [VAS] by the participant on a 100 mm visual analogue scale where higher scores indicate greater severity.
Awake Cough Frequency at Week 12 | Week 12
  Assessed using an ambulatory cough monitor
Percentage of Participants With >= 30 percent (%) Reduction From Baseline in 24-Hour Cough Frequency at Week 12 | Baseline, Week 12
  Assessed using an ambulatory cough monitor
Change from Baseline in the Leicester Cough Questionnaire (LCQ) Total Score at Week 12 | Baseline, Week 12
  The LCQ is a patient-reported quality of life (QOL) measure of chronic cough. The questionnaire consists of 19 items to which the patient responds on a 7-point Likert response scale (from 1 to 7). Each item assesses symptoms during cough and the impact of cough on 3 domains: physical, psychological, and social. Domain scores range from 1-7, and the total score ranges from 3 - 21; a higher score indicates a better quality of life.
Percentage of Participants With a >= 1.3-point Increase From Baseline in Leicester Cough Questionnaire (LCQ) Total Score at Week 12 | Baseline, Week 12
  The LCQ is a patient-reported quality of life (QOL) measure of chronic cough. The questionnaire consists of 19 items to which the patient responds on a 7-point Likert response scale (from 1 to 7). Each item assesses symptoms during cough and the impact of cough on 3 domains: physical, psychological, and social. Domain scores range from 1-7, and the total score ranges from 3 - 21; a higher score indicates a better quality of life.
Change from Baseline in the Chronic Cough Diary (CCD) Score at Week 12 | Baseline, Week 12
  The CCD is a participant-completed daily diary used to assess chronic cough. The CCD score ranges from 0 to 16, with a higher score indicating worse symptoms.
Percentage of Participants with CCD Response at Week 12 | Week 12
  Percentage of participants with CCD response will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (164):
- United States (60):
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Oak Lawn, Illinois
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Crowley, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Jersey City, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Little River, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Bellevue, Washington
  - GSK Investigational Site, Bellingham, Washington
- Argentina (10):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
  - GSK Investigational Site, Vicente López
- Belgium (7):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Roeselare
- Canada (14):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Victoriaville, Quebec
  - GSK Investigational Site, Burlington
- Colombia (2):
  - GSK Investigational Site, Floridablanca
  - GSK Investigational Site, Medellín
- France (7):
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
- Hungary (7):
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Hajdúnánás
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Püspökladány
- India (11):
  - GSK Investigational Site, Aurangabad
  - GSK Investigational Site, Bengaluru
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Kozhikode
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Rohtak
  - GSK Investigational Site, Thane
  - GSK Investigational Site, Ulhasnagar
- Israel (6):
  - GSK Investigational Site, Hadera
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
- Netherlands (7):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Uden
  - GSK Investigational Site, Zutphen
  - GSK Investigational Site, Zwolle
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Piaseczno
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Zawadzkie
- South Africa (6):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Durban
  - GSK Investigational Site, George
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
- Spain (9):
  - GSK Investigational Site, Alcobendas
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pozuelo de Alarcón
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (10):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Corby
  - GSK Investigational Site, Hayle
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
  - GSK Investigational Site, Northwood
  - GSK Investigational Site, Orpington
  - GSK Investigational Site, Shipley
  - GSK Investigational Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thach T, Dhanabalan K, Nandekar PP, Stauffer S, Heisler I, Alvarado S, Snyder J, Subramanian R. Mechanistic insights into the selective targeting of P2X3 receptor by camlipixant antagonist. J Biol Chem. 2025 Jan;301(1):108109. doi: 10.1016/j.jbc.2024.108109. Epub 2024 Dec 18. PMID 39706278